CLINICAL TRIAL: NCT07235696
Title: A Randomized Controlled Trial to Examine the Impact of a Game-based Intervention in Promoting Positive Affectivity and Enhancing Psychological Resilience
Brief Title: Game Intervention for Resilience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zhengxi Shao, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA250229
Record Dates: First submitted 2025-09-24; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Stress; Trauma Exposure; Resilience, Psychological; Major Life Stress
Keywords: Game-Based Intervention; Psychological Resilience; Major Life Stress; Positive Affectivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game-based intervention (Experimental)
  Interventions: Behavioral: Game-based Intervention
- Waitlist control (No Intervention)

INTERVENTIONS:
Behavioral: Game-based Intervention — This intervention is a two-week game-based program designed to enhance psychological resilience and positive affectivity in individuals who have experienced major life stress. The game incorporates emotionally engaging features such as reward mechanisms, adaptive challenge levels, and implicit emotion-regulation cues. Unlike traditional psychoeducation or mindfulness-based interventions, this program uses interactive gameplay to target affective and cognitive processes associated with resilience.
  Arms: Game-based intervention

SUMMARY:
The goal of this clinical trial is to learn if a game-based intervention can enhance psychological resilience and promote positive affectivity in adults who have experienced major life stress.

The main questions it aims to answer are:

* Does the game-based intervention improve positive affectivity and mental health compared to a waitlist control group immediately after the intervention and at 3-month follow-up?
* Are the mental health benefits of the game-based intervention mediated by improvements in positive affectivity over time?

Researchers will compare the game-based intervention to a waitlist control group to see if the game leads to better emotional and mental health outcomes.

Participants will:

* Be randomly assigned to either the game-based intervention group or the waitlist control group
* Engage with the assigned program for 10 days within two weeks
* Complete psychological assessments before and after the intervention, and again at 3-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* fluency in oral and written Cantonese or Mandarin;
* having experienced at least one major life stress in the recent 5 years (assessed by the Life Stress Index);
* normal or corrected-to-normal vision and hearing.

Exclusion Criteria:

* formal diagnosis of any major psychiatric illnesses or history of suicidal behaviour;
* major physical illness, neurological condition or traumatic brain injury;
* Intake of medication within the previous 6 months that may affect emotion or cognitive functions;
* pregnancy (for women);
* prior experience with any commercial computer repair simulation game.

Ages: 23 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Symptom-Checklist 90 (SCL-90) at Post-Assessment and 3-Month Follow-Up | Baseline, Post-Intervention (2 weeks), and 3-Month Follow-Up
  This outcome assesses changes in participants' psychological symptoms using the Symptom-Checklist 90 (SCL-90), a validated self-report instrument that measures a broad range of psychological problems and symptoms of psychopathology. Scores will be collected at baseline, immediately after the two-week intervention, and at 3-month follow-up to evaluate the effectiveness of the game-based intervention in improving mental health outcomes.

SECONDARY OUTCOMES:
Change from Baseline in the Positive Affect Assessed by Chinese Affect Scale (CAS) at Post-Assessment and 3-Month Follow-Up | Baseline, Post-Intervention (2 weeks), and 3-Month Follow-Up
  This outcome assesses changes in positive affect using the positive affect subscale of the Chinese Affect Scale (CAS). The measure will help determine whether the game-based intervention enhances emotional well-being.
Change from Baseline in Positive Refocusing Strategy Measured by the Cognitive Emotion Regulation Questionnaire (CERQ) at Post-Assessment and 3-Month Follow-Up | Baseline, Post-Intervention (2 weeks), and 3-Month Follow-Up
  This outcome evaluates changes in participants' use of positive refocusing as an emotion regulation strategy, measured by the corresponding subscale of the Cognitive Emotion Regulation Questionnaire (CERQ). The measure captures the tendency to redirect attention toward positive aspects during stressful experiences.
Change from Baseline in Positive Reframing Strategy Measured by the Brief COPE at Post-Assessment and 3-Month Follow-Up | Baseline, Post-Intervention (2 weeks), and 3-Month Follow-Up
  This outcome assesses changes in participants' use of positive reframing as a coping strategy, measured by the positive reframing subscale of the brief COPE inventory. This subscale reflects the ability to reinterpret stressful situations in a more positive light.
Change from Baseline in Mental Health Symptoms Assessed by Beck Depression Inventory-II (BDI-II) at Post-Assessment and 3-Month Follow-Up | Baseline, Post-Intervention (2 weeks), and 3-Month Follow-Up
  This outcome assesses changes in participants' psychological symptoms using the Symptom-Checklist 90 (SCL-90), a validated self-report instrument that measures a broad range of psychological problems and symptoms of psychopathology. Scores will be collected at baseline, immediately after the two-week intervention, and at 3-month follow-up to evaluate the effectiveness of the game-based intervention in improving mental health outcomes.
Change from Baseline in Reward Processing Assessed by Monetary Incentive Delay (MID) Task at Post-Assessment and 3-Month Follow-Up | Baseline, Post-Intervention (2 weeks), and 3-Month Follow-Up
  This outcome evaluates participants' behavioral responses to reward anticipation and motivated actions using the Monetary Incentive Delay (MID) Task. The task measures responses to reward, punishment, and neutral conditions, providing insight into the intervention's impact on reward-related brain function.
Change from Baseline in Cognitive Control Assessed by Color Stroop Task at Post-Assessment and 3-Month Follow-Up | Baseline, Post-Intervention (2 weeks), and 3-Month Follow-Up
  This outcome assesses participants' cognitive control and attentional regulation using the Color Stroop Task. Reaction time and accuracy will be measured to evaluate changes in executive functioning following the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No